CLINICAL TRIAL: NCT05565638
Title: PROlonged Nightly FASTing for Obesity Reduction and Prevention of Disease Prevention in Precursor Multiple Myeloma (PROFAST)
Brief Title: PROFAST Intervention in Precursor Multiple Myeloma
Acronym: PROFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Catherine Marinac, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-071; R21CA256644-01A1 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cancer Prevention; Weight Loss; Smoldering Waldenstrom Macroglobulinemia(WM); MGUS; Fasting; Multiple Myeloma
Keywords: Cancer prevention; Weight loss; Smoldering Waldenstrom Macroglobulinemia(WM); MGUS; Smoldering Multiple Myeloma; Prolonged nightly fasting; Multiple Myeloma
MeSH Terms: conditions — Weight Loss; Fasting; Multiple Myeloma; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PROLONGED FASTING INTERVENTION (Experimental): The prolonged nightly fasting (PROFAST) intervention involves gradually working up to a 14-hour fast during the nighttime hours. Participants will be supported by means of calls with a health coach during the first 4 weeks of the study. Participants will also be asked to use a text messaging platform to record their first and last meal of the day, and will receive personalized feedback based on the meal times they record via the text messaging system. The text messaging system will be used throughout the duration of the study.
  Interventions: Behavioral: Prolonged Fasting Intervention
- EDUCATION CONTROL (Active Comparator): For participants randomized to the control group, an introductory session with a health coach and educational information will be provided. Participants will also receive one email and one text message per week with tips on healthy living during the 4 months of the study
  Interventions: Behavioral: EDUCATION CONTROL

INTERVENTIONS:
Behavioral: Prolonged Fasting Intervention — promote a 14-hour fast during the nighttime hours
  Arms: PROLONGED FASTING INTERVENTION
Behavioral: EDUCATION CONTROL — introductory session with a health coach and educational information will be provided. Participants will also receive one email and one text message per week with tips on healthy living
  Arms: EDUCATION CONTROL

SUMMARY:
This is a 4-month randomized trial of a prolonged nightly fasting intervention (PROFAST) in 40 overweight and obese individuals with monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), and smoldering waldenstrom macroglobulinemia (SWM). The purpose of this study is to understand if fasting for a prolonged period of time during the nighttime hours is a strategy to prevent overweight and obese individuals from developing blood cancer.

Participants will be randomized into the following two groups:

* Group A: PROFAST intervention for 4 months
* Group B: Healthy Lifestyle Control group for 4 months

DETAILED DESCRIPTION:
The purpose of this research study is to learn if fasting for a prolonged period of time could be used in the future to help improve body composition and prevent blood cancer in overweight and obese individuals with MGUS, SMM, and SWM. Multiple myeloma is a cancer of the plasma cells, which is an important part of the immune system. Participants with active multiple myeloma generally require treatment. There are currently no approved therapies or prevention strategies for smoldering multiple myeloma or monoclonal gammopathy of undetermined significance.

The National Cancer Institute of the National Institutes of Health is supporting this research study by providing funding.

This research study is a 4-month randomized trial of prolonged nightly fasting (PROFAST). It is expected that about 40 people will take part in this research study. The total study duration is 4 months.

Participants in the study will be randomized, in equal numbers to either the nightly fasting intervention group or a control group.

* The prolonged nightly fasting (PROFAST) intervention involves gradually working up to a 14-hour fast during the nighttime hours. Participants will be supported by means of calls with a health coach during the first 4 weeks of the study. Participants will also be asked to use a text messaging platform to record their first and last meal of the day, and will receive personalized feedback based on the meal times via the text messaging system. The text messaging system will be used throughout the duration of the study.
* For participants randomized to the control group, an introductory session with a health coach and educational information will be provided. Participants will also receive one email and one text message per week with tips on healthy living during the 4 months of the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 25 kg/m2
* Documented diagnosis of MGUS or Smoldering MM(SMM) or Smoldering Waldenstrom Macroglobulinemia(WM) via EMR review. *note: please review case with PI or treating MD if diagnosis is uncertain.
* At least 18 years of age
* Currently fasting for <14 hours per night, as assessed using 24-hour food recalls
* Owns a cell phone and is comfortable sending and receiving text messages
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Diagnosis of overt MM or WM
* Patients diagnosed with another malignancy requiring active therapy
* Clinical diagnosis of diabetes, which may increase the risk of hypoglycemia with a prolonged fast. Note: patients with diabetes may enroll with consent from MD that manages their clinical care.
* Any other condition that, in the investigator's judgment, would contraindicate prolonged nightly fasting or otherwise interfere with participation in the trial, including night shift work, night eating syndrome, taking weight loss medication, or participation in another weight loss program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | baseline to 4-months
  assessed via whole body DXA scans

SECONDARY OUTCOMES:
M-Protein change by Serum Protein Electrophoresis and Serum Free Light Chain assay | baseline to 4-months
  Monoclonal (M-)proteins produced in excess by an abnormal clonal proliferation of plasma (MM) cells that can be measured in the serum using Serum Protein Electrophoresis (SPEP) and the Serum Free Light Chain Assay.
(M-)protein concentrations/light chains change by mass spectrometry | Baseline to 4-months
Changes in bone marrow adiposity | Baseline to 4-months
Changes in plasma metabolites measured by liquid chromatography-mass spectrometry | Baseline to 4-months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Marinac, Ph.D, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee DJ, O'Donnell EK, Raje N, Panaroni C, Redd R, Ligibel J, Sears DD, Nadeem O, Ghobrial IM, Marinac CR. Design and Rationale of Prolonged Nightly Fasting for Multiple Myeloma Prevention (PROFAST): Protocol for a Randomized Controlled Pilot Trial. JMIR Res Protoc. 2024 Mar 11;13:e51368. doi: 10.2196/51368. PMID 38466984